CLINICAL TRIAL: NCT01806272
Title: A Open,Randomized Phase II Trial Comparing Local Use of rhGM-CSF and Compound Vitamin B12 Solution to Compound Vitamin B12 Solution Alone Treating Chemoradiotherapy-induced Oral Mucositis in Patients With Primary Nasopharyngeal Carcinoma
Brief Title: Recombinant Human Granulocyte Macrophage Colony Stimulating Factor(rhGM-CSF) Treating Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei LUO (Other)
Responsible Party: Sponsor-Investigator, Wei LUO, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-12-01
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Nasopharyngeal Cancers
Keywords: rhGM-CSF; Oral Mucositis; Primary Nasopharyngeal Cancers; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Stomatitis | interventions — regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Local use of rhGM-CSF + Compound Vitamin B12 solution: The rhGM-CSF is prepared as a mouthwash solution,diluting 150μg in 100ml water(final concentration of 1.5μg/ml).Patient is instructed to use the solution five times daily.
  Compound Vitamin B12 solution 5ml being sprayed to mouth five times daily
  Radiotherapy: Intensity modulated radiation therapy(IMRT)
  Chemotherapy:Docetaxel or cisplatin weekly or cisplatin once every three weeks during radiotherapy.
  Interventions: Drug: rhGM-CSF; Drug: Compound Vitamin B12
- Arm B (Active Comparator): Compound Vitamin B12 solution 5ml being sprayed to mouth five times daily
  Radiotherapy: Intensity modulated radiation therapy(IMRT)
  Chemotherapy:Docetaxel or cisplatin weekly or cisplatin once every three weeks during radiotherapy.
  Interventions: Drug: Compound Vitamin B12

INTERVENTIONS:
Drug: rhGM-CSF — The rhGM-CSF is prepared as a mouthwash solution,diluting 150μg in 100ml water(final concentration of 1.5μg/ml).Patient is instructed to use the solution five times daily.
  Other Names: 特尔立
  Arms: Arm A
Drug: Compound Vitamin B12 — Compound Vitamin B12 solution 5ml being sprayed to mouth five times daily
  Other Names: 贯新克

SUMMARY:
This is a open,randomized phase II trial comparing effectiveness and safety of local use of rhGM-CSF and Compound Vitamin B12 to Compound Vitamin B12 solution alone treating oral mucositis in primary nasopharyngeal cancer. The main end point is the incidence of grade II and less oral mucositis at the end of treatment.The hypothesis of the study is that the local use of rhGM-CSF and Compound Vitamin B12 can decrease the incidence of grade III and more oral mucositis at the end of treatment compared to local use of Compound Vitamin B12 alone.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Grade II oral mucositis induced by chemoradiotherapy in patient with primary nasopharyngeal carcinoma.
2. Receiving 68-72 Gray of radiation dose.
3. Age between 18 and 65 years.
4. KPS≥70.
5. Patient who has given his/her written consent before any specific procedure of the protocol.

Exclusion Criteria:

1. Severe uncontrolled infection.
2. Pregnant or breast-feeding females.
3. Allergy to this medicine.
4. Diarrhea.

Outcome measures:

1. Grade of oral mucositis:NCI Common Terminology Criteria for Adverse Events v3.0, NCI CTCAE v3.0
2. Pain: WHO,Numerical Rating Scale(NRS)
3. Tumor response to chemoradiotherapy:Response Evaluation Criteria in Solid Tumors,RECIST1.1

ELIGIBILITY:
Inclusion Criteria:

1. Grade II oral mucositis induced by chemoradiotherapy in patient with primary nasopharyngeal carcinoma.
2. Receiving 68-72 Gray of radiation dose.
3. Age between 18 and 65 years.
4. KPS≥70.
5. Patient who has given his/her written consent before any specific procedure of the protocol.

Exclusion Criteria:

1. Severe uncontrolled infection.
2. Pregnant or breast-feeding females.
3. Allergy to this medicine.
4. Diarrhea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade II and less oral mucositis at the end of treatment | 7 weeks
  Using the criteria of NCI CTCAE v3.0

SECONDARY OUTCOMES:
Pain | 12 weeks
  Cumulative incidence and time of different grade,using the criteria of WHO,NRS
Cumulative incidence and time of grade III and more oral mucositis | 7 weeks
  Using the criteria of NCI CTCAE v3.0
Dysphagia | 12 weeks
  Cumulative incidence and time of different grade,using NCI CTCAE v3.0
Tumor response to chemoradiotherapy | 12 weeks
  Using the criteria of Response Evaluation Criteria in Solid Tumors1.1(RECIST1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Wei LUO, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China